CLINICAL TRIAL: NCT00445159
Title: An Investigator Initiated Eight Week Two Center Open-Label Pilot Study of the Tolerability and Safety of Oral UT-15C (Treprostinil Diethanolamine)SR Tablets in Patients With Critical Limb Ischemia (CLI) and Ischemic Rest Pain
Brief Title: UT-15C SR in the Treatment of Critical Limb Ischemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern Arizona Vascular Institute (Other)
Collaborators: Southern Illinois University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UT-15C
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2007-03-08 (Estimated); Status verified 2007-03

CONDITIONS: Critical Limb Ischemia
Keywords: UT-15C SR, Peripheral Vascular Disease, treprostinil
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Vascular Diseases | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: UT-15C SR (treprostinil diethanolamine) 1mg oral tablets

SUMMARY:
This study will evaluate UT-15C sustained release tablets in subjects experiencing ischemic lower limb rest pain related to advanced peripheral arterial disease. Rest pain is one of the primary management issues of severe arterial occlusive disease and may lead to amputation when the pain becomes intolerable and unresponsive to narcotic analgesia. Rest pain also impacts the quality of sleep and mobility with frequent interruptions in sleep and decreased mobility. Treprostinil sodium (Remodulin®) has been studies in several small open-label studies and has been shown to be safe as well as an effective agent for ischemic rest pain when given by subcutaneous or intravenous delivery. However, these forms of administration have patient convenience limitations, including the need for an infusion device and associated pain at the site of infusion with subcutaneous delivery. UT-15C may allow patients suffering from CLI to benefit from the simplicity of an oral dosage form

DETAILED DESCRIPTION:
This study is an eight week, two center, open-label study assessing the tolerability, safety, and efficacy of oral UT-15C sustained release tablets in subjects with CLI and ischemic lower limb rest pain, with or without an ischemic wound present. Conventional therapy should be continued without changes over the course of the study for all subjects.

Group 1: The first ten subjects to enroll in the study will be assigned to receive an initial dose of 1mg. The dose will be titrated upward every seven days, depending on tolerability, to a maximum dose of 4mg/day .

Group 2: The last ten subjects to enroll in the study will be assigned to receive an initial dose of 1mg. The dose will be titrated upward every seven days, depending on tolerability to a maximum dose of 8 mg/day .

ELIGIBILITY:
Inclusion Criteria:

1. Have an ankle systolic pressure ≤ 60 mm/Hg OR ABI ≤ 0.60 OR toe systolic pressure ≤ 60 mm/Hg OR an arteriogram showing at least one level of occlusion of lower extremity arteries.
2. Have been taking analgesics to control ischemic rest pain for at least two weeks at Baseline.
3. Have signed an appropriate consent for participation in this study.
4. If female, be physiologically incapable of childbearing or practicing acceptable methods of birth c

Exclusion Criteria:

1. Have had a vascular surgery or other vascular procedure to treat their CLI within 30 days prior to study entry.
2. Have a planned or scheduled vascular surgery or endovascular procedure.
3. Be currently taking any investigational drugs for CLI.
4. Have received prostaglandins such as PGE1, epoprostenol (Flolan®), or any other prostacyclin (PGI2) or prostacyclin analog in the past 30 days.
5. Be hemodynamically unstable or have acute renal failure, cardiac failure or pulmonary failure.
6. Have a diagnosis of Stage IVb (Fontaine) or Stage 6 (Rutherford scale) Critical Limb Ischemia due to documented peripheral arterial disease
7. Have an unhealed incision(s) from a toe or transmetatarsal amputation at Baseline.
8. Have any wound with significant gangrene or exposed tendons.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-11

PRIMARY OUTCOMES:
To assess the tolerability and safety of UT-15C tablets in subjects with critical limb ischemia (CLI) and ischemic rest pain

SECONDARY OUTCOMES:
To assess the effect of UT-15C on the following disease symptoms associated with CLI:
ž Ischemic rest pain
ž Sleep interference
ž Ambulatory status
ž Ischemic wound healing (if applicable)
To obtain peak and trough treprostinil plasma levels in CLI subjects

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Johnson, MD, Principal Investigator — Southern Illinois University; Scott S Berman, MD, Principal Investigator — Southern Arizona Vascular Institute
Locations (2):
- United States (2):
  - Southern Arizona Vascular Institute, Tucson, Arizona
  - Southern Illinois University School of Medicine, Springfield, Illinois